CLINICAL TRIAL: NCT06385730
Title: Neoadjuvant PD-1 Blockade (Toripalimab) Monotherapy for Elderly Patients With Locally Advanced Resectable Esophageal Squamous Cell Carcinoma: a Phase II Trial
Brief Title: Neoadjuvant PD-1 Blockade for Elderly Esophageal Squamous Cell Carcinoma (BLESS)
Acronym: BLESS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Li, Chief of Department of Esophageal Surgery, Shanghai Chest Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCE2401
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer, immunotherapy, elderly patients
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoadjuvant anti-PD-1 (Experimental): Drug: Immunotherapy Patients will receive the neoadjuvant immunotherapy with toripalimab followed by the esophagectomy.
  Interventions: Drug: neoadjuvant anti-PD-1
- neoadjuvant anti-PD-1 with LDRT (Experimental): Drug: Immunotherapy Patients will receive the neoadjuvant low-dose radiotherapy plus immunotherapy with toripalimab followed by the esophagectomy.
  Interventions: Drug: neoadjuvant anti-PD-1 with LDRT

INTERVENTIONS:
Drug: neoadjuvant anti-PD-1 — PD-1 inhibitor (toripalimab) 240mg, day 1，every 3 weeks, 2 cycles. Postoperative adjuvant treatment: according to the recommendations of the guidelines and the investigators
  Arms: neoadjuvant anti-PD-1
Drug: neoadjuvant anti-PD-1 with LDRT — Radiotherapy: low-dose radiotherapy (LDRT), gross target volume (GTV), DT: 1Gy (day1), 1Gy (day2), every 3 weeks, 2 cycles.
  PD-1 inhibitor (toripalimab) 240mg, day 3，every 3 weeks, 2 cycles. Postoperative adjuvant treatment: according to the recommendations of the guidelines and the investigators
  Arms: neoadjuvant anti-PD-1 with LDRT

SUMMARY:
The investigators will conduct a prospective phase 2 study to evaluate the efficacy and safety of neoadjuvant PD-1 blockade monotherapy with toripalimab in elderly patients with locally advanced resectable esophageal squamous cell carcinoma (ESCC).

DETAILED DESCRIPTION:
The incidence and mortality rates of esophageal cancer both rapidly increase after the age of 40 to 50 and peak after the age of 70 to 80. Clinical studies have shown that over 50% of esophageal cancer patients are diagnosed at an advanced local stage. Currently, the standard treatment recommended by guidelines for locally advanced esophageal cance is neoadjuvant chemoradiotherapy or chemotherapy. However, the phase III randomized controlled trials upon which these recommendations are based did not include patients over 75 years old. Therefore, for elderly patients aged over 75 with locally advanced esophageal cancer, there remains a lack of high-level evidence-based optimal neoadjuvant treatment strategies in clinical practice.

In Japan, neoadjuvant chemotherapy combined with surgery is the standard treatment for locally advanced esophageal cancer. A retrospective analysis (PMID: 35837977) conducted at 85 esophageal cancer centers certified by the Japan Esophageal Society examined patients with esophageal squamous cell carcinoma who received neoadjuvant CF (cisplatin + 5-fluorouracil) or intensified neoadjuvant DCF (docetaxel + cisplatin + 5-fluorouracil) regimens. The study results showed that the survival benefit of intensified neoadjuvant DCF was limited to patients aged ≤75 years. In patients older than 75 years, no survival advantage of intensified neoadjuvant DCF was observed, and the incidence of postoperative pneumonia was higher. The study suggested that elderly patients may not tolerate the toxic side effects of intensified neoadjuvant DCF triplet therapy. The high-intensity neoadjuvant triplet chemotherapy increased the incidence of postoperative complications in esophageal cancer, possibly offsetting the survival benefit in terms of tumor eradication.

A phase 1 trial conducted in 2023 (PMID: 37488287) demonstrated that neoadjuvant single-agent immunotherapy (atezolizumab) for locally advanced resectable esophageal squamous cell carcinoma is safe, with no Grade 3 or higher adverse reactions. The primary pathological response rate was 24%, with a complete pathological response rate of 8%. The 2-year overall survival rate was 92%, and the 2-year recurrence-free survival rate reached 100%. When compared with a historical control study (CMISG1701 study), the 2-year recurrence-free survival rate and 2-year overall survival rate with neoadjuvant single-agent immunotherapy were significantly higher, showing a statistically significant improvement compared to both standard neoadjuvant chemoradiotherapy (61% vs. 69%) and standard neoadjuvant chemotherapy (63% vs. 67%).

Based on (1) clinical evidence indicating higher adverse reactions and limited benefits of high-intensity neoadjuvant treatment regimens in elderly esophageal squamous cell carcinoma patients and (2) the potential advantages of neoadjuvant single-agent immunotherapy over standard neoadjuvant chemoradiotherapy or chemotherapy in terms of safety and survival benefits, this trial reasonably proposes a scientific research proposal-to explore the efficacy and safety of neoadjuvant immunotherapy monotherapy in elderly (aged over 75) patients with locally advanced thoracic esophageal squamous cell carcinoma under conditions of reduced combination therapy and decreased adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects signed the informed consent and volunteered to participate in the study.
2. Esophageal squamous cell carcinoma confirmed by histology or cytology.
3. Thoracic esophageal squamous cell carcinoma confirmed by CT or pet-CT, which is classified as T1N1-3M0 or T2-3N0-3M0 (M1 lymph node metastasis confined to the supraclavicular lymph nodes) (AJCC 8th).
4. Expect to have R0 resection
5. In age >75.
6. ECOG PS: 0~1.
7. Have not received any anti-tumor treatment for esophageal cancer in the past, including radiotherapy, chemotherapy, surgery, etc.
8. No contraindications to surgery.
9. Has sufficient organ function including (1) Blood routine: NE≥1.5×109/L; PLT≥100×109/L; HGB≥90 g/L (2)Comprehensive Metabolic Panel: bilirubin≤ 1.5×ULN; ALT≤2.5×ULN; AST≤2.5×ULN; sCr≤1.5×ULN or CrCl≥50 mL/min（Cocheroft-Gault) (3) Coagulation function: INR≤1.5.
10. Women of childbearing age must undergo a serological pregnancy test within 72 hrs before first administration. Women of childbearing age, or male subjects with childbearing age female partners, must take contraceptive measures from the first dose to five months after last administration.
11. Good compliance, willing to comply with follow-up schedules.

Exclusion Criteria:

1.Subjects have received or are receiving any of:

1. anti-tumor interventions such as radiotherapy, chemotherapy, immunotherapy or other medictions.
2. Received systemic corticosteroid therapy (prednisone equivalence> 10mg/d) or other immunosuppressive agents within the first 2 weeks prior to the first administration.
3. live vaccine within 4 weeks before the first administration.

2. Cancer related exclusion criteria

1. other cancers instead of ESCC
2. non-recetable or metastatic ESCC
3. not comply with T1N1-3M0 or T2-3N0-3M0 (AJCC 8th).
4. Subjects with other malignant tumors within 5 years before the first administration, but subjects with cervical carcinoma in situ, skin basal cell carcinoma, skin squamous cell carcinoma, and localized prostate cancer received radical surgery in situ that have received radical treatment and do not need other treatment can be included).

3. Other criteria Subjects have uncontrolled cardiovascular diseases, such as 1) heart failure ≥ NYHA class 2, 2) unstable angina 3) myocardial infarction within 1 year; 4) supraventricular or ventricular arrthymia that needs treatment Subjects with any known active autoimmune disease Pregnant or breastfeeding female Presence of allergy or hypersensitivity to investigational medications HIV positive or active hepatitis B (HbsAg positive and HBV-DNA ≥2000 IU/ml or ≥ 104 copies/mL) or active hepatitis C (HCV antibody positive) or active tuberculosis Investigators assessed there might be other factors that cause subjects to withdrawl.

Min Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
MPR rate | Through the study completion, an average of 12 months
  A major pathological response rate (MPR) is defined as the proportion of residual living tumor cells in the post-surgery specimen within the tumor bed being less than or equal to 10%

SECONDARY OUTCOMES:
pCR rate | Through the study completion, an average of 12 months
  The primary endpoint is a pCR rate, which is defined as the absence of any remaining tumor cells in both the main tumor and the nearby lymph nodes (ypT0N0) as per the AJCC 8th Edition TRG scoring system
Adverse events and treatment-related adverse events | Through the study completion, an average of 12 months
  Including adverse events and complications. Incidence of adverse events using CTCAE 5.0; grade 3 treatment-related adverse events and higher-grade will be reported
R0 resection rate | Through the study completion, an average of 12 months
  A R0 resection rate is defined as the rate of complete tumor removal with negative resection margin microscopically
Objective Response rate | Through the study completion, an average of 12 months
  objective response (according to the Response Evaluation Criteria In Solid Tumors, version 1.1)
Event-free survival (EFS) | Through the study completion, an average of 12 months
  An event-free survival (EFS) is defined as the duration from the start of treatment until disease progression/recurrence or death from any cause, whichever occurs first.
Overall survival (OS) | Through the study completion, an average of 24 months
  Overall survival (OS) is defined as the time from treatment to death, regardless of disease recurrence
Correlation between potential biomarkers and tumor response | Through the study completion, an average of 36 months
  Tumor microenvironment (assessed by genomic sequencing) will be correlated with tumor response

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yin J, Yuan J, Li Y, Fang Y, Wang R, Jiao H, Tang H, Zhang S, Lin S, Su F, Gu J, Jiang T, Lin D, Huang Z, Du C, Wu K, Tan L, Zhou Q. Neoadjuvant adebrelimab in locally advanced resectable esophageal squamous cell carcinoma: a phase 1b trial. Nat Med. 2023 Aug;29(8):2068-2078. doi: 10.1038/s41591-023-02469-3. Epub 2023 Jul 24. PMID 37488287
- [Background] Matsuda S, Kitagawa Y, Takemura R, Okui J, Okamura A, Kawakubo H, Muto M, Kakeji Y, Takeuchi H, Watanabe M, Doki Y. Real-world Evaluation of the Efficacy of Neoadjuvant DCF Over CF in Esophageal Squamous Cell Carcinoma: Propensity Score-matched Analysis From 85 Authorized Institutes for Esophageal Cancer in Japan. Ann Surg. 2023 Jul 1;278(1):e35-e42. doi: 10.1097/SLA.0000000000005533. Epub 2022 Jul 15. PMID 35837977
- [Background] Yang Y, Zhu L, Cheng Y, Liu Z, Cai X, Shao J, Zhang M, Liu J, Sun Y, Li Y, Yi J, Yu B, Jiang H, Chen H, Yang H, Tan L, Li Z. Three-arm phase II trial comparing camrelizumab plus chemotherapy versus camrelizumab plus chemoradiation versus chemoradiation as preoperative treatment for locally advanced esophageal squamous cell carcinoma (NICE-2 Study). BMC Cancer. 2022 May 6;22(1):506. doi: 10.1186/s12885-022-09573-6. PMID 35524205